CLINICAL TRIAL: NCT03238651
Title: A Phase 1, Open-label Study of TAK-659 as a Single Agent in Adult East Asian Patients With Non-Hodgkin Lymphoma
Brief Title: A Study of TAK-659 as a Single Agent in Adult East Asian Participants With Non-Hodgkin Lymphoma (NHL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of the study by the sponsor due to business decision.
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C34007; U1111-1186-6838 (Registry Identifier: WHO)
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Follicular, Marginal Zone
Keywords: Drug therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — TAK-659

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Part Schedule A: TAK-659 60 mg in Cohort 1 (Experimental): TAK-659, tablet, orally, once daily, in a 28-day treatment cycle for up to 12 months or until disease progression or unacceptable toxicity, with a starting dose of 60 milligram (mg) in Cohort 1. Dose escalation will follow a standard 3+3 schema . If 60 mg, once daily is safe and tolerable, then the dose will be escalated to 80 mg, once daily and subsequently in 20 mg increments until MTD and/or RP2D is determined. Based on emerging safety, tolerability, PK data, a lower dose will be permitted.
  Interventions: Drug: TAK-659
- Dose Escalation Part Schedule B: TAK-659 80 mg in Cohort 1 (Experimental): TAK-659, tablet, orally, once daily as 7 days on and 7 days off treatment (dosing on 7 days followed by 7 days of rest) in a 28-day treatment cycle for up to 12 months or until disease progression or unacceptable toxicity, with a starting dose of 80 mg in Cohort 1. Dose escalation will follow a standard 3+3 schema. An alternative intermittent regimen may be evaluated if deemed necessary per the emerging data.
  Interventions: Drug: TAK-659
- Expansion Part: TAK-659 MTD/RP2D (Experimental): TAK-659, tablet, orally, once daily, in a 28-day treatment cycle until disease progression or unacceptable toxicity in participants with follicular lymphoma (FL) or marginal zone lymphoma (MZL) who are relapsed and/or refractory. Dose and dosing schedule for this part will be MTD/RP2D determined from results of dose escalation part.
  Interventions: Drug: TAK-659

INTERVENTIONS:
Drug: TAK-659 — TAK-659 Tablets.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of TAK-659 when administered in East Asian participants with NHL who do not have an effective standard treatment available and to characterize the plasma and urine pharmacokinetic (PK) of TAK-659 in East Asian participants with NHL.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-659. TAK-659 is being tested to treat people who have NHL or people who have relapsed and/or refractory NHL. This study will assess the safety, tolerability, PK, and preliminary efficacy of single-agent TAK-659 in East Asian participants with NHL.

The study will enroll approximately 33 to 47 participants, including at least 6 Japanese at RP2D dose level. Participants will be assigned to one of the following treatment groups:

Dose Escalation Part: TAK-659 Expansion Part: TAK-659 RP2D

This multi-center trial will be conducted in Japan and Republic of Korea. The maximum duration of participation in dose escalation part of the study is up to 12 months, unless in the opinion of the investigator and sponsor the participant would derive benefit from continued therapy beyond 12 months. In expansion part, participants who stop treatment for any other reason other than PD will continue to have PFS follow-up at the site every 2 months from the last dose of study drug up to 6 months or until PD. Participants will be followed 28 days after last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurs first, for a follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. To be enrolled to the dose escalation part, participants must have histologically or cytologically confirmed diagnosis of NHL for which no effective standard treatment is available.
2. To be enrolled in the expansion part, participants must meet the following criteria:

   1. Must have pathologically confirmed FL (Grade 1, 2, or 3A) or MZL.
   2. Relapsed and/or refractory to >=2 prior lines of chemotherapy based on standard of care that include at least 1 anti-CD20-based regimen, as well as alkylating agents (example cyclophosphamide or bendamustine).
   3. Participants must be ineligible for or refusal to hematopoietic stem cell transplant.
   4. If the participants have relapsed or progressed after achieving a response (defined as CR or PR), documented, investigator-assessed relapse or progression after the last treatment is required.
3. Measurable disease per IWG 2007 criteria.
4. Eastern Cooperative Oncology Group performance status score of 0 or 1.
5. Life expectancy of longer than 3 months.
6. Adequate organ function, including the following:

   1. Bone marrow reserve: absolute neutrophil count >=1,000 per cubic millimeter (/mm^3), platelet count >=75,000/mm^3 (>=50,000/mm^3 for participants with bone marrow involvement), and hemoglobin >=8 gram per deciliter (g/dL) (red blood cell [RBC] and platelet transfusion allowed >=14 days before assessment).
   2. Hepatic function: total bilirubin less than or equal to (<=) 1.5*the upper limit of the normal range (ULN); alanine aminotransferase and aspartate aminotransferase <=2.5*ULN.
   3. Renal function: creatinine clearance >=60 milliliter per minute (mL/min) either as estimated by the Cockcroft-Gault equation.

Exclusion Criteria:

1. Central nervous system (CNS) lymphoma; active brain or leptomeningeal metastases as indicated by positive cytology from lumbar puncture or computed tomography (CT)/magnetic resonance imaging (MRI) by local assessment.
2. Systemic anticancer treatment (including investigational agents) less than 3 weeks before the first dose of study treatment (<=4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agent; <=8 weeks for cell-based therapy or anti-tumor vaccine).
3. Radiotherapy less than (<) 3 weeks before the first dose of study treatment. If prior radiotherapy occurred <4 to 6 weeks before the study start, as radiated lesions cannot be reliably assessed by fluoro-2-deoxy-D-glucose (FDG)-positron emission tomography (PET), nonradiated target lesions are required for eligibility.
4. Prior autologous stem cell transplant (ASCT) within 6 months or prior ASCT at any time without full hematopoietic recovery before Cycle 1 Day 1, or allogeneic stem cell transplant at any time.
5. Any clinically significant comorbidities, such as uncontrolled pulmonary disease (example, severe chronic obstructive pulmonary disease with hypoxemia, interstitial lung disease, radiation induced lung injury), known impaired cardiac function or clinically significant cardiac disease, active CNS disease, or any other condition that could, in the opinion of the investigator, compromise the participant's safety and participation in the study per protocol.
6. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659.
7. Use or consumption of any of the following substances:

Received medications, supplements, or food/beverages that are P-glycoprotein (P-gp) inhibitors or inducers or strong cytochrome P450 (CYP) 3A inhibitors or inducers within a certain time frame prior to the first dose of study drug. Depending on the substance, the washout period for P-gp inhibitors or inducers or strong CYP3A inhibitors or inducers will be either 7 days or 5 times the half-life (half-life is related to the time required for elimination from the body). The washout period for grapefruit containing food or beverages is 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Japan (2):
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Japan and South Korea from 1 August 2017 to 17 August 2020.
Pre-assignment Details: Participants with non-Hodgkin lymphoma (NHL) were enrolled in 1 of the 2 treatment schedules in the Dose Escalation Part to receive TAK-659: Dosing Schedule A and Dosing Schedule B. Dose Expansion part was not initiated and the data for secondary outcome measures was not analyzed due to early termination of the study by the sponsor due to business decision.
Groups:
- Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg: TAK-659 40 milligram (mg), tablet, orally, once daily, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
- Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg: TAK-659 60 mg, tablet, orally, once daily, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
- Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg: TAK-659 80 mg, tablet, orally, once daily, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
- Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg: TAK-659 80 mg, tablet, orally, once daily as 7 days on and 7 days off treatment (dosing on 7 days followed by 7 days of rest) in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
- Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg: TAK-659 100 mg, tablet, orally, once daily as 7 days on and 7 days off treatment (dosing on 7 days followed by 7 days of rest) in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
Period: Overall Study
Arm/Group | Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Started | 3 | 6 | 4 | 3 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 4 | 3 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 2 | 2 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Groups:
- Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg: TAK-659 40 mg, tablet, orally, once daily, in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg | Total
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.50) | 64.5 (19.46) | 63.3 (8.92) | 65.7 (2.89) | 67.0 | 64.9 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 1 | 5
  Male | 3 | 5 | 2 | 2 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 4 | 3 | 1 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 4 | 3 | 1 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 1 | 4 | 2 | 1 | 0 | 8
  Korea, Republic Of | 2 | 2 | 2 | 2 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: From first dose of study drug up to 28 days after the last dose of study drug or before the start of subsequent anticancer therapy (up to Cycle 31) (Cycle length =28 days)
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg: TAK-659 40 mg, tablet, orally, once daily, in a 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal due to other reasons.
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
percentage of participants | 100 | 100 | 100 | 100 | 100

2. Primary Outcome: Percentage of Participants With Grade 3 or Higher TEAEs
Description: TEAEs were graded as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. As per the NCI-CTCAE, Grade 1 (mild, asymptomatic or mild symptoms); Grade 2 (moderate, minimal, local or noninvasive intervention indicated); Grade 3 (severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (life-threatening consequences, urgent intervention indicated); Grade 5 (death related to adverse event [AE]).
Time Frame: as for outcome 1
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
percentage of participants | 66.7 | 100 | 100 | 100 | 0

3. Primary Outcome: Percentage of Participants With Serious TEAEs
Time Frame: as for outcome 1
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
percentage of participants | 0 | 100 | 75 | 33.3 | 100

4. Primary Outcome: Dose Escalation Part: Percentage of Participants With Dose-limiting Toxicities (DLTs) During Cycle 1
Description: DLT was evaluated as per NCI-CTCAE, v4.03 and defined as any of the following events occurring during Cycle 1 that were considered by the investigator to be possibly related to therapy: Grade 4 neutropenia unresolved to less than or equal to (<=) Grade 1 or baseline for more than 7 days in the absence of growth factor support; greater than or equal to (>=) Grade 3 neutropenia with fever and/or infection;Grade 4 thrombocytopenia unresolved to <=Grade 1 or baseline for more than 7 days; >=Grade 3 thrombocytopenia with clinically significant bleeding; Grade >=3 nonhematologic toxicity except for treated >=Grade 3 nausea and/or emesis and diarrhea resolved to less than (<) Grade 3 within 3 days, Grade 3 fatigue <=72 hours, isolated asymptomatic >=Grade 3 laboratory abnormalities resolved to <=Grade 1 or baseline in <=7 days;received <75% of planned doses of study drug in Cycle 1;TAK-659-related >=Grade 2 nonhematologic toxicities that required dose reduction or discontinuation of therapy.
Time Frame: Cycle 1 (Cycle length =28 days)
Population: DLT-evaluable analysis set included participants who met the minimum treatment and safety evaluation requirements of the study or who experienced a DLT during Cycle 1. As planned, this outcome measure was analyzed and reported for dose escalation part only.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
percentage of participants | 0 | 16.7 | 50 | 0 | 0

5. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to TEAEs
Time Frame: as for outcome 1
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
percentage of participants | 33.3 | 50 | 50 | 0 | 0

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-659 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The pharmacokinetic (PK) analysis set included participants who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
nanogram per milliliter (ng/mL) | 93.86 (62.88) | 127.65 (22.39) | 214.50 (74.67) | 216.00 (18.01) | 297.00

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-659 on Cycle 1 Day 7 (Dosing Schedule B) and Cycle 1 Day 15 (Dosing Schedule A)
Time Frame: Cycle 1 Day 7 (Dosing Schedule B) and Day 15 (Dosing Schedule A): pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 2 | 3 | 1
ng/mL | 121.18 (39.57) | 130.23 (62.95) | 308.29 (53.67) | 339.42 (29.96) | 329.00

8. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-659 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
hours | 1.97 [1.0 to 3.0] | 3.01 [1.9 to 4.0] | 2.00 [0.5 to 3.0] | 2.05 [0.5 to 2.7] | 2.00 [2.0 to 2.0]

9. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-659 on Cycle 1 Day 7 (Dosing Schedule B) and Cycle 1 Day 15 (Dosing Schedule A)
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 2 | 3 | 1
hours | 3.00 [0.5 to 3.1] | 3.01 [0.0 to 4.1] | 2.25 [0.5 to 4.0] | 2.00 [0.9 to 2.0] | 1.00 [1.0 to 1.0]

10. Primary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-659 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg: TAK-659 40 mg, tablet, orally, once daily, in a 28-days treatment cycle disease progression, unacceptable toxicity, or withdrawal due to other reasons.
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 1
hour*nanogram per milliliter (h*ng/mL) | 587.2534 (22.2886) | 1207.6554 (26.3167) | 1742.7394 (39.3327) | 1899.2508 (15.1827) | 1828.4544

11. Primary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-659 on Cycle 1 Day 7 (Dosing Schedule B) and Day 15 (Dosing Schedule A)
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 0
h*ng/mL | 1114.2391 (1.1927) | 2016.8000 (21.3348) | 3502.3513 (25.0980) | 3349.4133 (12.2891) |

12. Primary Outcome: CLR: Renal Clearance for TAK-659 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15: pre-dose and at multiple time points (up to 8 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure. CLR data was planned to be collected and analyzed for both of the Dosing Schedule A and B arms. However, urine sample was not collected in Dosing Schedule B due to administrative reasons. Therefore, data was not analyzed and reported for schedule B arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Dose Escalation Part, Schedule Dosing A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
Number analyzed (Participants) | 3 | 6 | 2 | 0 | 0
liter per hour (L/h) | 6.7303 (49.0441) | 8.4185 (114.6567) | 9.4059 (22.3501) |  |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were adverse events that started from first dose of study drug up to 28 days after the last dose of study drug or before the start of subsequent anticancer therapy (up to Cycle 31) (Cycle length =28 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/4 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 6/6 | 3/4 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg (N=3) | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg (N=6) | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg (N=4) | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg (N=3) | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg (N=1)
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Part, Dosing Schedule A: TAK-659 40 mg (N=3) | Dose Escalation Part, Dosing Schedule A: TAK-659 60 mg (N=6) | Dose Escalation Part, Dosing Schedule A: TAK-659 80 mg (N=4) | Dose Escalation Part, Dosing Schedule B: TAK-659 80 mg (N=3) | Dose Escalation Part, Dosing Schedule B: TAK-659 100 mg (N=1)
Pyrexia (General disorders) | 0 | 1 | 3 | 1 | 1
Face oedema (General disorders) | 0 | 3 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 4 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 4 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 3 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03238651/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03238651/SAP_001.pdf